CLINICAL TRIAL: NCT06677411
Title: Annual Fluctuation of Vitamin D Nutritional Status in Students and Its Association with the Occurrence of Inflammation, Depressive States, and Cognitive Abilities
Brief Title: Vitamin D Status Fluctuations Over One Academic Year in Students
Status: Active, not recruiting | Type: Observational
Sponsor: Poznan University of Life Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: VITDstud
Record Dates: First submitted 2024-09-03; First posted 2024-11-06 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-06

CONDITIONS: Vitamin D Deficiency
MeSH Terms: conditions — Vitamin D Deficiency

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- University students
  Interventions: Other: Observention of vitamin D

INTERVENTIONS:
Other: Observention of vitamin D — It is an observational study

SUMMARY:
The main objective of the study is to assess changes in the concentration of vitamin D metabolite in serum throughout the academic year and to examine its relationship with the occurrence of inflammation indicators, dietary habits, nutritional status, severity of depressive states, and cognitive abilities in a group of students. An additional objective will be to assess the relationship between the genotype in the CYP2R1 gene and the concentration of 25(OH) vitamin D.

ELIGIBILITY:
Inclusion Criteria:

* no chronic diseases
* student status
* age 18-30 years

Exclusion Criteria:

* chronic diseases (related to malabsorption, kidney and liver diseases)
* not active student status
* age <18 and >30 years

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Study population includes students of both sexes at the age of 18-30 years who agree to participate and attend all four study meetings over one academic year. The participants should be in good health condition.
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Vitamin D concentration | 01.10.2024-01.10.2025
  Measurement of 25(OH) vitamin D in serum at four points over an academic year

SECONDARY OUTCOMES:
Inflammation status measured with CRP | 01.10.2024-01.10.2025
Depressive symptoms | 01.10.2024-01.10.2025
  The magnitude of depressive symptoms over an academic year
Cognitive functions | 01.10.2024-01.10.2025
Body composition | 01.10.2024-01.10.2025
Dietary intake of vitamin D | 01.10.2024-01.10.2025
CYP2R1 genotype | 01.10.2024-01.10.2025

CONTACTS AND LOCATIONS:
Overall Officials: Emilia Zawieja, PhD, Principal Investigator — Poznan University of Life Sciences
Locations (2):
- Poland (2):
  - Poznan University of Life Sciences, Poznan, Wielkopolska
  - Poznan University of Life Sciences, Poznan